CLINICAL TRIAL: NCT01283022
Title: A Multicenter, Open-Label, Phase II Study of the 200 mcg Misoprostol Vaginal Insert (MVI 200) to Obtain Pharmacokinetics in Women at Term Gestation (The MVI-PK Study)
Brief Title: Pharmacokinetic (PK) Study of the 200 Microgram (mcg) Misoprostol Vaginal Insert (MVI 200) in Women at Term Gestation (The MVI-PK Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Miso-Obs-205
Record Dates: First submitted 2011-01-20; First posted 2011-01-25 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Cervical Ripening; Induction of Labor
Keywords: Pharmacokinetics; Misoprostol Vaginal Insert; Induction of labor; Cervical Ripening; Rate of Cesarean section

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MVI 200 (Experimental): MVI 200 mcg vaginal insert
  Interventions: Drug: MVI 200

INTERVENTIONS:
Drug: MVI 200 — Dose reservoir of 200 mcg of misoprostol in a hydrogel polymer vaginal insert within a retrieval system. The MVI 200 will be kept in place for up to 24 hours or will be removed earlier if one of the following occur: onset of active labor, intrapartum adverse event necessitating discontinuation of the study drug, other reasons including maternal request.
  Other Names: Misopess (TM); Misodel (R)

SUMMARY:
The purpose of this study is to determine the pharmacokinetics (PK) of misoprostol acid for the MVI 200 in women requiring cervical ripening and induction of labor.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent;
* Pregnant women at ≥ 36 weeks 0 days inclusive gestation;
* Women aged 18 years or older;
* Candidate for pharmacologic induction of labor;
* Single, live vertex fetus;
* Baseline modified Bishop score ≤ 4;
* Parity ≤ 3 (parity is defined as one or more births live or dead after 24 weeks gestation);
* Body Mass Index (BMI) ≤ 50 at the time of entry to the study.

Exclusion Criteria:

* Women with hemoglobin level < 10.0 grams per deciliter (g/dL) (confirmed within one week of study drug insertion);
* Women in active labor;
* Presence of uterine or cervical scar or uterine abnormality e.g., bicornate uterus. Biopsies, including cone biopsy of the cervix, are permitted;
* Administration of oxytocin or any cervical ripening or labor inducing agents (including mechanical methods) or a tocolytic drug within 7 days prior to enrollment. Magnesium sulfate is permitted if prescribed as treatment for pre-eclampsia or gestational hypertension;
* Severe pre-eclampsia marked by Hemolytic anemia, Elevated Liver enzymes, Low Platelet count (HELLP) syndrome, other end-organ affliction or Central Nervous System (CNS) findings other than mild headache;
* Fetal malpresentation;
* Diagnosed congenital anomalies, not including polydactyly;
* Any evidence of fetal compromise at baseline (e.g., non-reassuring fetal heart rate pattern or meconium staining);
* Amnioinfusion or other treatment of non-reassuring fetal status at any time prior to the induction attempt;
* Ruptured membranes ≥ 48 hours prior to the start of treatment;
* Suspected chorioamnionitis;
* Fever (oral or aural temperature > 37.5°C);
* Any condition in which vaginal delivery is contraindicated e.g., placenta previa or any unexplained genital bleeding at any time after 24 weeks during this pregnancy;
* Known or suspected allergy to misoprostol, other prostaglandins or any of the excipients;
* Any condition urgently requiring delivery;
* Unable to comply with the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Huntington Memorial Hospital, Pasadena, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant women who required to be induced were recruited at 1 site in the US
Groups:
- MVI 200: MVI 200 : Dose reservoir of 200 mcg of misoprostol in a hydrogel polymer vaginal insert within a retrieval system. The MVI 200 will be kept in place for up to 24 hours or will be removed earlier if one of the following occur: onset of active labor, intrapartum adverse event necessitating discontinuation of the study drug, other reasons including maternal request.
Period: Overall Study
Arm/Group | MVI 200
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MVI 200
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (6.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of Misoprostol After Insertion
Description: The timepoints over which the pharmacokinetic measurements were assessed, and deemed as accurate and appropriate, were as follows: 0 hours (baseline), 0.5,1, 2, 4, 6, 8, 10 and 14 hours after insertion of the study drug, immediately prior to removal of the study drug and 0.5 and 1 hour after removal of the study drug. The 10 hour and 14 hour blood samples were obtained if the subject still had the study drug in place at those timepoints.
Time Frame: From study drug insertion up to 1 hour post study drug removal.
Population: The pharmacokinetic (PK) analysis included all 24 subjects from the Intention-to-Treat (ITT) population.
Measure: Median (Standard Deviation); unit: hours
Arm/Group | MVI 200
Number analyzed (Participants) | 24
hours | 4 (2.09)

2. Secondary Outcome: Rate of Adverse Events.
Description: All adverse events were rated by the Investigator as mild, moderate or severe and classified as having no relationship, possible relationship or a probable relationship to the study drug. These assessments were deemed as accurate and appropriate for the reporting of all serious and non serious adverse events.
Time Frame: From study drug administration to hospital discharge (approximately 48-72 hours).
Population: The percentage of subjects with adverse events are presented for the Intrapartum (before delivery), postpartum (maternal) and neonatal periods.
Measure: Number; unit: percentage of participants
Arm/Group | MVI 200
Number analyzed (Participants) | 24
percentage of participants
  Subjects with Intrapartum Adverse Events | 66.7
  Subjects with Maternal Postpartum Adverse Events | 8.3
  Subjects with Neonatal Adverse Events | 50.0

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Misoprostol up to 1 Hour Post Study Drug Removal
Description: as for outcome 1
Time Frame: From study drug insertion up to 1 hour post study drug removal
Population: The pharmacokinetic (PK) analysis included all 24 subjects from the Intention-to-Treat (ITT) population.
Measure: Median (Standard Deviation); unit: pg/mL
Arm/Group | MVI 200
Number analyzed (Participants) | 24
pg/mL | 45.8 (25.7)

ADVERSE EVENTS:
Time Frame: All adverse events were followed until resolution or for at least 30 days after discontinuation of study drug, whichever occurred first.
Description: All adverse events occurring to the maternal-fetal unit (pre-delivery/ intrapartum), the mother (postpartum) or the neonate were recorded. Adverse events that resulted in a cesarean delivery were reported as serious adverse events as they were medically significant events that routinely prolonged the duration of hospitalization.
Arm/Group | MVI 200
Serious Adverse Events (participants affected / at risk) | 5/24
Other Adverse Events (participants affected / at risk) | 16/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVI 200 (N=24)
Cryptorchism * (Congenital, familial and genetic disorders) | 1 (1) — * Neonatal Event
Hydrocele * (Congenital, familial and genetic disorders) | 1 (1) — * Neonatal Event
Abnormal labour affecting foetus + (Pregnancy, puerperium and perinatal conditions) | 1 (1) — + Intrapartum Event
Foetal heart rate disorder + (Pregnancy, puerperium and perinatal conditions) | 2 (2) — + Intrapartum Event
Infantile apnoeic attack * (Respiratory, thoracic and mediastinal disorders) | 1 (1) — * Neonatal Event
Neonatal respiratory distress syndrome * (Respiratory, thoracic and mediastinal disorders) | 1 (1) — * Neonatal Event
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVI 200 (N=24)
Abnormal labour affecting foetus + (Pregnancy, puerperium and perinatal conditions) | 2 (3) — + Intrapartum Event
Arrested labour + (Pregnancy, puerperium and perinatal conditions) | 5 (5) — + Intrapartum Event
Foetal heart rate disorder + (Pregnancy, puerperium and perinatal conditions) | 5 (5) — + Intrapartum Event
Meconium in amniotic fluid + (Pregnancy, puerperium and perinatal conditions) | 5 (5) — + Intrapartum Event
Umbilical cord around neck * (Pregnancy, puerperium and perinatal conditions) | 4 (4) — * Neonatal Event
Uterine contractions abnormal + (Pregnancy, puerperium and perinatal conditions) | 2 (2) — + Intrapartum Event
Hypotension + (Vascular disorders) | 3 (3) — + Intrapartum Event
Apgar score low * (Investigations) | 2 (2) — * Neonatal Event
Caput succedaneum * (Pregnancy, puerperium and perinatal conditions) | 2 (2) — * Neonatal Event
Cephalohaematoma * (Pregnancy, puerperium and perinatal conditions) | 2 (2) — * Neonatal Event
Infection prophylaxis * (Surgical and medical procedures) | 3 (3) — * Neonatal Event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any abstract,presentation or manuscript proposed for publication must be submitted to the Sponsor for review at least 30 days prior to submission for any meeting or journal.If deemed necessary by the Sponsor for protection of proprietary information prior to patent filing,the Investigator agrees to a further delay of 60 days before any presentation or publication is submitted.Publications must be in a form that does not reveal technical information that is considered confidential or proprietary.